CLINICAL TRIAL: NCT05543408
Title: Long COVID-19 Syndrome in Primary Care: A Novel Protocol of Exercise Intervention "CON-VIDA Clinical Trial"
Acronym: CON-VIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Lucia Sagarra, PhD, Universidad San Jorge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Universidad San Jorge
Record Dates: First submitted 2022-09-15; First posted 2022-09-16 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Long COVID; Post-COVID-19 Syndrome
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXERCISE (Experimental)
  Interventions: Behavioral: EXERCISE
- CONTROL (No Intervention)

INTERVENTIONS:
Behavioral: EXERCISE — individualized, progressive, exercise program
  Arms: EXERCISE

SUMMARY:
This is a randomized controlled trial of the efficacy of an individualized, progressive, exercise program (strength, cardiovascular, and breathing exercises) in recovering people from the post-COVID-19 syndrome (i.e., patients who present symptoms >12 weeks once the acute phase of the disease is over).

DETAILED DESCRIPTION:
This is a randomized controlled trial of the efficacy of an individualized, progressive, exercise program (strength, cardiovascular, and breathing exercises) in recovering people from the post-COVID-19 syndrome (i.e., patients who present symptoms >12 weeks once the acute phase of the disease is over). The primary objective of the study is to evaluate the clinical efficacy and safety of a tailored exercise-based treatment relative to the control arm in improving the subject clinical status in both ambulatory and hospitalized post-COVID-19 syndrome patients. The main novelty of this trial compared to other exercise-based interventions is the development and proof of concept of a progressively, levelled exercise regime for people with physical activity intolerance and fatigue symptoms.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years of age.
* Persistent symptoms of COVID >3 months of duration since infection.
* Have no medical contraindications incompatible with the practice of exercise.
* Do not meet the general 2020 recommendations for physical activity established by the World Health Organization2 (i.e., at least 150-300 minutes of moderate-intensity aerobic physical activity; or at least 75-150 minutes of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week).
* Provide signed informed consent.

Exclusion Criteria:

* Presence of uncontrolled serious medical illness.
* Presence of any medical, psychological or social problem that could seriously interfere with the patient's participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Lower Limb Strength: 30 s Sit-to-Stand test | Baseline to 8 weeks
  The test starts with the participant seated on a chair (43.2 cm), arms crossed at the wrists and held against the chest. From this position, participants will conduct as much as sit-to-stand repetitions, as fast as possible, during 30 s
Change in Lower Limb Strength: 5 times Sit-to-Stand Test | Baseline to 8 weeks
  Participants will have to sit and stand 5 times (as quickly as possible) from a chair (43.2 cm), arms crossed at the wrists and held against the chest. Time will be register.
Change in Handgrip Strength | Baseline to 8 weeks
  Start by holding the instrument in the testing hand. Squeeze the dynamometer handle as hard as possible to obtain peak force values.
Chance in upper limbs strength: Arm Curl Biceps | Baseline to 8 weeks
  The subject sits on chair, holding the weight in the hand using suitcase grip, with the arm in a vertically downward position beside the chair. Curl the arm up through a full range of motion, gradually returns to the starting position. The arm must be fully bent and then fully straightened at the elbow. The aim of this test is to do as many arm curl as possible in 30 seconds.
Change in Balance: Flamingo Balance Test | Baseline to 8 weeks
  Number of seconds keeping balance with one foot on the floor and the other resting on the opposite ankle (maximum 60 s)
Change in walking speed: Brisk Walking Test | Baseline to 8 weeks
  Number of seconds required to walk 30 m.
Change in cardiovascular fitness: 6-Minute Walk Test | Baseline to 8 weeks
  Number of meters that can be walked in 6 min around 30 m track.
Change in pulmonary function: Inspiratory and Expiratory Pressures | Baseline to 8 weeks
  The maximal inspiratory pressure (MIP) and Maximum Expiratory Pressure (MEP) reflects the respiratory muscles ability to generate force during a short quasi-static contraction.
  MIP and MEP measurements are conducted with a manometer that measures mouth pressure and these depend on the motivation and co-ordination of the patient.
  Procedures:
  * MIP: from tidal breathing the patient slowly exhales as deeply as possible. During expiration the measurement is started manually. The shutter will be set as soon as the patient starts to breathe in. Now the patient is asked to inspire as fast and as powerful as possible against the shutter. The maximal inspiratory pressure will be reached after about 0.5-1 s.
  * MEP: from tidal breathing the patient slowly breathes in as deeply as possible. The shutter will be closed with expiration onset. Now the patient is asked to expire as fast and as powerful as possible against the shutter.
Change in pulmonary function: Peak flow Test | Baseline to 8 weeks
  Peak expiratory flow measurement (peak flow) is a simple measure of the maximal flow rate that can be achieved during forceful expiration following full inspiration.
  First, the patient should reset the meter by sliding the marker all the way to zero on the scale. While sitting or standing up straight, the patient should take in a full, deep breath. The mouthpiece is then placed in the patient's mouth followed by a single, fast, forceful expiration. The marker will slide outward on the numbered scale, indicating the peak expiratory flow rate for that attempt.

SECONDARY OUTCOMES:
Body Composition | Baseline to 8 weeks
  Bio-Electrical Impedance Analysis (BIA) with 200 kg maximum capacity and 50 g error margin (TANITA BC-418MA, Tanita Corp., Tokyo, Japan).The meassurement includes: body weight (kg) body fat mass, the percentage of body fat (BF%) and the fat-free mass (FFM). Body mass index (BMI) will be calculated dividing weight (kg) by squared height (m2).
Change in Quality of Life-SF-36 | Baseline to 8 weeks
  The SF-36 is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Change in The International Physical Activity Questionnaire (IPAQ) | Baseline to 8 weeks
  The International Physical Activity Questionnaires (IPAQ) comprises a set of 4 questionnaires.
  Long (5 activity domains asked independently) and short (4 generic items) versions for use by either telephone or self-administered methods are available. The purpose of the questionnaires is to provide common instruments that can be used to obtain internationally comparable data on health-related physical activity.
Change in Modified Medical Research Council dyspnea scale (mMRC) | Baseline to 8 weeks
  The mMRC Dyspnea Scale is used to assess the degree of baseline functional disability due to dyspnea in patients with respiratory problems. The mMRC breathlessness scale ranges from grade 0 to 4 (low to high).
Change in Modified Fatigue Impact Scale (MFIS) | Baseline to 8 weeks
  The MFIS measures the impact fatigue takes on a patient's daily life. It consists of 21 items divided into 3 subdivision containing 9 physical items , 10 cognitive items and 2 psychosocial. All the items are rated from 0-4 .
  The sum of all the questions are calculated where 84 is the highest score. Highest the score means higher the impact of fatigue in daily living.
Change in Hospital Anxiety and Depression Scale (HADS) | Baseline to 8 weeks
  HADS is a fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Change in the short form of the DePaul Symptom Questionnaire (DSQ-SF) | Baseline to 8 weeks
  The short for of the DSQ-SF is a self-report measure of demographic characteristics, myalgic encephalomyelitis and chronic fatigue syndrome symptomatology, and medical, occupational, and social history.
Change in the Insommia Severity Index (ISI) | Baseline to 8 weeks
  The ISI is composed of seven items that evaluate the severity of sleep disturbance during the past 2 week
  * The first three items assess the severity of difficulties with falling sleep, maintaining sleep, and early morning awakening.
  The last four items capture satisfaction with the current sleep patte, interference with daily functioning, noticeability of impairment, and degree of distress caused by the sleep problem.
  The scores of each of the seven items range from 0 to 4 (0 = none; 4 = very severe), and a total score can be calculated by summing the seven items, giving a range from 0 to 28, with higher scores indicating greater insomnia severity. Total scores are interpreted as 0-7, absence of insomnia; 8-14, sub-threshold insomnia; 15-21, moderate insomnia; 22-28, severe insomnia.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucia Sagarra-Romero, Zaragoza, Spain